CLINICAL TRIAL: NCT04308070
Title: Acute Hemostasis Following the Use of the AQUABEAM® System for the Treatment of Benign Prostatic Hyperplasia III
Acronym: AHAIII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: PROCEPT BioRobotics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TP0148
Record Dates: First submitted 2017-10-04; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Benign Prostatic Hyperplasia
Keywords: Image-guided; BPH; Aquablation; AQUABEAM; LUTS; Tissue resection; Robotics
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Catheter without Hemostatic Agent Following Aquablation (Experimental): AQUABEAM System followed by catheter without hemostatic agent
  Interventions: Device: AQUABEAM System followed by catheter without hemostatic agent
- Catheter with Hemostatic Agent Following Aquablation (Experimental): AQUABEAM System followed by catheter with hemostatic agent
  Interventions: Device: AQUABEAM System followed by catheter with hemostatic agent

INTERVENTIONS:
Device: AQUABEAM System followed by catheter without hemostatic agent — The AquaBeam system delivers a high-pressure saline stream under precise electromechanical control and live ultrasound guidance to ablate prostatic glandular tissue without the production of heat. The physician uses ultrasound imaging to plan the treatment contour and depth to define the treatment region. The physician will use balloon catheter to achieve hemostasis post-Aquablation procedure.
  Arms: Catheter without Hemostatic Agent Following Aquablation
Device: AQUABEAM System followed by catheter with hemostatic agent — The AquaBeam system delivers a high-pressure saline stream under precise electromechanical control and live ultrasound guidance to ablate prostatic glandular tissue without the production of heat. The physician uses ultrasound imaging to plan the treatment contour and depth to define the treatment region. The physician will use balloon catheter with hemostatic agent to achieve hemostasis post-Aquablation procedure.
  Arms: Catheter with Hemostatic Agent Following Aquablation

SUMMARY:
A dual-arm prospective, interventional clinical trial to evaluate the safety and performance of obtaining hemostasis with catheters along with the use or absence of a hemostatic agent following treatment with the AQUABEAM System.

DETAILED DESCRIPTION:
PROCEPT BioRobotics has developed the AQUABEAM, a personalized image-guided waterjet resection system that utilizes a high-pressure saline stream to resect and remove prostate tissue in males suffering from LUTS due to BPH. The primary objective of this study is to evaluate the safety and performance of obtaining hemostasis using balloon catheters with and without hemostatic agents following prostate resection using AQUABEAM for the treatment of LUTS resulting from BPH. Up to 50 participants will be included in the trial at one clinical study site. All patients will be followed up for 3 months for safety assessment prior to study exit. The trial is a dual-arm prospective, interventional clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Male
* BPH symptoms

Exclusion Criteria:

* Serious concurrent medical conditions

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2017-07-18 (Actual); Primary Completion 2018-03-22 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Number of subjects that do not require a transfusion and do not return to the operating room for hematuria management within 7 days following the index procedure. | 7 days post-op
  Adequate hemostasis post-Aquablation with the use of a urinary catheter and / or delivery of a hemostatic agent, measured by the number of subjects that, within 7 days following the index procedure, do not require a transfusion and do not return to the operating room for hematuria management.

CONTACTS AND LOCATIONS:
Locations (1):
- Muljibhai Patel Urological Hospital, Nadiād, Gujarat, India

IPD SHARING:
Plan to Share IPD: Undecided